CLINICAL TRIAL: NCT03889314
Title: The DEtermining Statin Intolerance FOr Rosuvastatin (DESIFOR) Trial
Acronym: DESIFOR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: DESIFOR
Record Dates: First submitted 2019-03-15; First posted 2019-03-26 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Cardiovascular Risk Factor; Cardiovascular Diseases; Adverse Effect
Keywords: Statin Therapy; Prevention; High ASCVD Risk
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Patients will serve as their own controls in this study whereby they will receive randomly allocated 28-day packets of statin and placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rosuvastatin 20mg (Experimental): Each participant will receive a 3 month randomly allocated supply of this medication preceded by a 7 day wash-out period.
  Interventions: Drug: Rosuvastatin 20mg
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- No Treatment (No Intervention): 7 day wash-out period between months

INTERVENTIONS:
Drug: Rosuvastatin 20mg — Statin Therapy
  Arms: Rosuvastatin 20mg
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will enroll patients who previously were not able to tolerate being on a statin medication due to muscle-related side effects. Research has shown that many people who have muscle symptoms on statin therapy do not experience the same side effects if they try it again later. This study is part of a larger effort to:

* See how common it is for patients to still be intolerant of statin medication after trying it a second time; and
* For those patients who do tolerate being on a statin after trying it a second time, see how common it is for them to still be taking the statin 3 months after completing the main part of the study.

Patients who agree to participate will be given a 5 month randomly allocated supply of statin and placebo and track their symptoms weekly.

DETAILED DESCRIPTION:
This study is a single center, double-blinded randomized controlled trial for patients eligible for statin therapy by current guidelines, but not on statin therapy due to a history of statin intolerance. Patients will be provided a "DESIFOR" kit which includes 5 randomly allocated 4-week blister packs of capsules containing either 20mg of rosuvastatin or placebo. While blinded to treatment, patients will document the severity of musculoskeletal symptoms every week using a numerical scale. The primary endpoint will be the difference between the mean musculoskeletal symptom score while randomized to statin therapy compared to the mean score while on placebo. After completion of the study, the results will be unblinded and reviewed at a 6 month follow-up visit with the patient and, for patients with symptoms found to not correlate with statin therapy, a trial of non-blinded statin therapy over the next 3 months will be recommended. This study will serve as a pilot study to determine the feasibility and potential benefits of a larger multicenter trial with similar aims.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 21-75 years old
* Statin eligible according to the 2013 ACC/AHA cholesterol guidelines, including individuals with:

  * Known ASCVD
  * Diabetes
  * LDL-C > 190mg/dl
  * 10-year ASCVD risk >7.5%
* Statin intolerant

  * Defined by discontinuation of at least 2 separate statins due to potential musculoskeletal side effects

Exclusion Criteria:

* Women who are pregnant, nursing or attempting to become pregnant.
* Individuals deemed to be at very high CVD risk and therefore appropriate for a PCSK9 inhibitor including:

  * Individuals with familial hypercholesterolemia with markedly elevated LDL-C levels
  * Individuals with known ASCVD and recurrent events
  * Individuals who are not otherwise clinically indicated to take 20mg rosuvastatin
* Individuals who experienced severe reactions in the past, including:

  * Rhabdomyolysis
  * Severe myositis
  * Anaphylaxis

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal intolerance (as documented in study assessments) | 6 months
  Prevalence of musculoskeletal intolerance between the groups, defined by a lack of statistical difference in the mean musculoskeletal symptom score while on statin therapy compared to placebo, in patients previously identified as statin intolerant.

SECONDARY OUTCOMES:
Statin Utilization | 3 months
  Number of individuals taking statins 3 months post study

CONTACTS AND LOCATIONS:
Overall Officials: Michael Miedema, MD, Principal Investigator — Minneapolis Heart Institute Foundation
Locations (1):
- Minneapolis Heart Institute Foundation, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No